CLINICAL TRIAL: NCT03025620
Title: Investigation of the Relationship Between Alpha-linolenic Acid and Arterial, Biochemical, Biological Parameters in Older Persons With History of Cardiovascular Events and/or Moderate Cognitive Impairment
Brief Title: Dietary Intake of Alpha-linolenic Acid in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Elevage (Unknown); ITERG (Industry); SAINT HUBERT (Unknown); TERRES UNIVIA (Unknown); TERRES INOVIA (Unknown)
Responsible Party: Principal Investigator, Fathi Driss, Doctor, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Alphalinolenage
Record Dates: First submitted 2017-01-10; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Diseases; Inflammation; Metabolism Disorder, Lipid
Keywords: Alphalinolenic acid; Lipid cardiovascular risk factors; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Lipid Metabolism Disorders | interventions — Rapeseed Oil; alpha-Linolenic Acid; Sunflower Oil; Linoleic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sunflower arm (Placebo Comparator): Participants were supplied with the usual diet of the hospital, daily enriched with 17.5g fat as follows during 42 days: 10 g of sunflower oil (with a high content in linoleic acid) were added into the dinner soup and 7.5g delivered through a 12.5g portion of margarine made with sunflower oil (60% fat) that replaced butter on the breakfast toasts.
  Interventions: Dietary Supplement: Sunflower oil
- Rapeseed arm (Active Comparator): Participants were supplied with the usual diet of the hospital, daily enriched with 17.5g fat as follows during 42 days: 10 g of rapeseed oil (with a high content in alpha-linolenic acid) were added into the dinner soup and 7.5g delivered through a 12.5g portion of margarine made with rapeseed oil (60% fat) that replaced butter on the breakfast toasts.
  Interventions: Dietary Supplement: Rapeseed oil

INTERVENTIONS:
Dietary Supplement: Rapeseed oil — Active comparator arm : Dietary Supplement: rapeseed oil supplementation (10g per day) and margarine with a high level of alpha-linolenic acid (12.5g per day) during 42 days.
  Other Names: Alpha-linolenic acid
  Arms: Rapeseed arm
Dietary Supplement: Sunflower oil — Placebo comparator arm : Dietary Supplement: sunflower oil supplementation (10g per day) and margarine with a high level of inoleic acid (12.5g per day) during 42 days.
  Other Names: Linoleic acid
  Arms: Sunflower arm

SUMMARY:
The purpose of this study is to evaluate the antiatherogenic and anti-inflammatory potential of an adequate intake of alpha-linolenic acid in elderly.

DETAILED DESCRIPTION:
There is growing evidence that diets high in long chain n-3 polyunsaturated fatty acids (PUFA) decrease the risk of fatal ischemic heart disease.Both epidemiologic studies and clinical trials demonstrate substantial cardioprotective effects of alpha linolenic acid (ALA) from vegetable oils.However, little is known about the relation of the dietary intake of ALA with ischemic heart disease among older adults.In this study, elderly volunteers will be asked to ingest a supplement of a vegetable oil providing 1g of ALA, or an equivalent amount of linoleic acid as sunflower oil, for a diet period of 6 weeks.Serum samples will be collected before the dietary intervention and 6 weeks later.Plasma biomarkers of inflammatory, lipid cardiovascular risk factors and serum and red cell membrane fatty acid composition will be determined on all samples.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients over 65 years old exhibiting clinical indices of cardiovascular disease
* Male or female
* Subjects who were hospitalized in the Geriatric Unit of the Emile Roux Hospital (AP-HP)
* MMSE (Mini Mental State Examination)score > or = 15
* Supervision available for study medication
* Able to ingest oral diet

Exclusion Criteria:

* Patients unable to understand the objectives of the dietary intervention
* Patients in paliative care
* Patients receiving supplement diets

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-11; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effects of diet supplementation on fatty acid composition in serum and red cell membrane phospholipids, at the end of dietary period | 6 weeks
  Blood samples have been done at the beginning and at the end of the dietary period. Fatty acids analyses of the red cells and serum have been performed by GC method.

SECONDARY OUTCOMES:
Pulse wave velocity (PWV) | 6 weeks
  Pulse wave velocity values have been performed at the beginning and the end of the dietary period.
  The purpose was to evaluate the relationship between PWV and dietary intakes of ALA.
Others | 6 weeks
  ApoB ApoA1 Oxydative parameters (ie CRP) Lp(a)

CONTACTS AND LOCATIONS:
Overall Officials: olivier henry, MD, Principal Investigator — Assistance Publique de Paris. Hopital Emile Roux
Locations (1):
- hopital Emile Roux, Limeil-Brévannes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giallauria F, Vigorito C, Tramarin R, Fattirolli F, Ambrosetti M, De Feo S, Griffo R, Riccio C, Piepoli M; ISYDE-2008 Investigators of the Italian Association for Cardiovascular Prevention, Rehabilitation, and Prevention. Cardiac rehabilitation in very old patients: data from the Italian Survey on Cardiac Rehabilitation-2008 (ISYDE-2008)--official report of the Italian Association for Cardiovascular Prevention, Rehabilitation, and Epidemiology. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1353-61. doi: 10.1093/gerona/glq138. Epub 2010 Jul 28. PMID 20667934
- [Background] Rodriguez-Leyva D, Dupasquier CM, McCullough R, Pierce GN. The cardiovascular effects of flaxseed and its omega-3 fatty acid, alpha-linolenic acid. Can J Cardiol. 2010 Nov;26(9):489-96. doi: 10.1016/s0828-282x(10)70455-4. PMID 21076723
- [Background] Salva A, Corman B, Andrieu S, Salas J, Vellas B; International Association Of Gerontology/International Academy Of Nutrition And Aging Task Force. Minimum data set for nutritional intervention studies in elderly people. J Gerontol A Biol Sci Med Sci. 2004 Jul;59(7):724-9. doi: 10.1093/gerona/59.7.m724. PMID 15304539
- [Background] Bischoff HA, Staehelin HB, Willett WC. The effect of undernutrition in the development of frailty in older persons. J Gerontol A Biol Sci Med Sci. 2006 Jun;61(6):585-9. doi: 10.1093/gerona/61.6.585. No abstract available. PMID 16799140
- [Background] Abbatecola AM, Cherubini A, Guralnik JM, Andres Lacueva C, Ruggiero C, Maggio M, Bandinelli S, Paolisso G, Ferrucci L. Plasma polyunsaturated fatty acids and age-related physical performance decline. Rejuvenation Res. 2009 Feb;12(1):25-32. doi: 10.1089/rej.2008.0799. PMID 19196012